CLINICAL TRIAL: NCT01517945
Title: Attention and Interpretation Modification (AIM) for Fear of Cancer Recurrence: An Intervention Development Study
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Brown University (Other); Weill Medical College of Cornell University (Other); Johns Hopkins University (Other); Mclean Hospital (Other); University of Southern California (Other); The New School for Social Research (Other)
Responsible Party: Sponsor
Other Study IDs: 11-204
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Rare Cancer
Keywords: Survivors; Quality of Life; Questionnaire; 11-204; Rare Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — salvia
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Breast cancer survivors and Rare cancer survivors: This is a Cycle for Survival and Center for Translational Science Center (CTSC)-funded intervention development and pilot clinical trial of a psychosocial intervention to address fear of cancer recurrence in breast cancer survivors (BCS) and rare cancer survivors (RCS). BCS form the largest survivor cohort of any cancer, with approximately 2.5 million living in the United States. About 50 percent of people with cancer have a rare cancer. Even though they account for about half of all cancer diagnoses when combined, research aimed at supporting RCS is sparse, leaving RCS with limited support after treatment.
  Interventions: Behavioral: AIM materials and assessments

INTERVENTIONS:
Behavioral: AIM materials and assessments — Phase 1 (complete) - dev of AIM materials targeting fear of cancer recurrence in BCS (n = 10).
  Phase 2 (complete) - randomized, single-blind, placebo-controlled, proof-of-concept pilot trial.
  Phase 3:
  * Part 1 of Phase 3 (complete) - dev of of iThrive app for BCS
  * Part 2 of Phase 3 (complete) - usability testing by observing navigation with BCS in a laboratory setting
  * Part 3 of Phase 3 - acceptability of iThrive will be assessed through a small RCT (n=30)
  Phase 4:
  * Part 1 of Phase 4 (complete) - dev of iThrive app for RCS
  * Part 2 of Phase 4 (complete) - usability testing completed by observing navigation with RCS remotely
  * Part 3 of Phase 4 - acceptability of iThrive will be assessed through a small RCT (n=90)
  For Phases 3 and 4, Part 3: We will work with participants to ensure that sessions are completed over < 12 weeks if unavoidable delays occur. A follow-up session will be scheduled 3 months after completion of the last session.
  Other Names: In situations where there are unanticipated and unavoidable session delays, we; will work with the participants to ensure that all sessions are completed over; no more than 12 weeks A follow-up session will be scheduled 3 months as far; back as 2 weeks before and as far out as 6 weeks after) after the completion; of session 8.

SUMMARY:
The purpose of this study is to test, customize, and personalize a mobile app-based intervention program in order to help rare and breast cancer survivors cope with fears of cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

Phases 1 & 2:

* Breast cancer survivors
* Hx of early-stage breast cancer (DCIS and Stages I, II and III)as recorded in the medical record at MSK or by self-report or by outside correspondence, including a study checklist signed by a physician for patients outside of MSK.
* ≥ 3 months post completion of breast cancer treatment (may be on hormone therapy, such as tamoxifen) with no history of recurrence or metastasis as confirmed by the medical record at MSK, self- report or by outside correspondence
* Age 18 or older
* Able to read and speak English
* An overall fear index score of ≥ 3.0 on the CARS
* If taking medication for mood, anxiety, depression, thoughts, sensory experiences such as hallucinations, or sleep, stable and consistent enough in dosage and use of that medication so as to not result in a clinically significant change as determined by the study PI/co-PI or confirmed by reports in the medical record at MSK or by self-report or by outside correspondence, including a study checklist signed by a physician for patients outside of MSK
* If in non-CBT psychotherapy, stable for at least 8 weeks
* Access to a computer or willingness to come to MSK to complete intervention sessions 2-8 and the 3-month follow-up assessment, if no personal computer.
* For Part 2 only, did not participate in Part 1

Phase 3, Part 1 and 2:

* Hx of early-stage breast cancer (DCIS and Stages I, II, and III) as recorded in the medical record at MSK or by self-report or by outside correspondence, including a study checklist signed by a physician for patients outside of MSK
* Completion of breast cancer treatment (may be on hormone therapy, such as tamoxifen) with no history of recurrence or metastasis as confirmed by the medical record at MSK, by self-report, or by outside correspondence
* Age 18 or older
* English fluency: self-report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* Score of >/= 12 on the 8-item Cancer Worry Scale
* Score of >/= 2 SDs below the mean on the euro-QOL-Short Form
* Uses an iOS mobile device (may be an iPad)
* If taking medication for mood, anxiety, depression, thoughts, sensory experiences such as hallucinations, or sleep, stable for at least 8 weeks and consistent enough in dosage and use of that medication so as to not result in a clinically significant change as determined by the study PI/co-PI or confirmed by reports in the medical record at MSK or by self-report or by outside correspondence, including a study checklist signed by a physician for patients outside of MSK.

Phase 3, Part 3:

* Hx of early-stage breast cancer (DCIS and Stages I, II, and III) with no history of metastasis as per EMR, by self-report, or by outside correspondence.
* Completion of breast cancer treatment (may be on hormone therapy, such as tamoxifen, or on maintenance medication) as per the EMR or self-report.
* Age 18 or older as per the EMR or self-report.
* English fluency: Self-report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well"
* Score ≥ 9 on the 6-item Cancer Worry Scale (CWS: this score was found to be optimal to screen for high FCR across cancer types)
* Score of > 2 SDs below the mean on the Neuro-QOL-Short Form
* Uses an iOS mobile device (may be an iPad) as per self-report.
* If taking medication for mood, anxiety, depression, thoughts, sensory experiences such as hallucinations, or sleep, stable for at least 8 weeks and consistent enough in dosage and use of that medication so as to not result in a clinically significant change as determined by the study PI/co-PI or confirmed by the EMR or by self-report or by outside correspondence including a study checklist signed by a physician for patients outside of MSK
* Must reside in the United States.

Phase 4, Parts 2 and 3:

* Hx of early stage (Stages 0, I, II, and III) rare melanoma subtypes (e.g., acral, uveal) and skin (excluding keratinocyte cancers, e.g., basal and squamous cell), gynecological, long-term adult, pediatric rare liquid cancer (in remission only) or other rare cancer per the EMR, by self-report, or by outside correspondence.
* Age 18 or older, as per the EMR or self-report.
* English fluency: Self-report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* Score ≥ 9 on the 6-item Cancer Worry Scale (CWS; this score was found to be optimal to screen for high FCR across cancer types)
* Score of >2 SDs below the mean on the Neuro-QOL - Short Form
* Uses an iOS mobile device (may be an iPad) as per self-report.
* If taking medication for mood, anxiety, depression, thoughts, sensory experiences such as hallucinations, or sleep, stable for at least 8 weeks and consistent enough in dosage and use of that medication so as to not result in a clinically significant change as determined by the study PI/co-PI or confirmed by the EMR or by self-report or by outside correspondence, including a study checklist signed by a physician for patients outside of MSK
* Completed active treatment (can be on hormonal therapy or on maintenance medication) as per the EMR or self-report.
* Must reside in the United States.

Exclusion Criteria:

Phases 1 & 2:

* Evidence of or treatment for a second primary of cancer EXCEPT basal or squamous cell carcinoma of the skin as confirmed by the EMR, by self-report, or by outside correspondence
* Significant psychiatric or cognitive disturbance sufficient, to preclude providing informed consent or participating in the interventions (i.e., acute psychiatric symptoms which require individual treatment) as determined by the study PI/co-PI or confirmed by the EMR or by self-report or by outside correspondence
* Current participation in cognitive-behavioral therapy (CBT), as confirmed by either self-report* or the EMR, also targets cognitive biases.

Phase 3:

* Evidence of or treatment for a second primary cancer EXCEPT basal or squamous cell carcinoma of the skin as confirmed by the medical record at MSK, by self-report, or by outside correspondence
* Metastatic disease
* Score of </= SDs below the mean on the Neuro-QOL-Short Form or other indicators of significant cognitive impairment of psychiatric disturbance that, in the PI's judgment, precludes participation; and currently receiving cognitive-behavioral therapy.

Phase 4:

* Metastatic disease as per the EMR or self-report.
* Score of ≤ 2 SDs below mean of the Neuro-QoL- Short Form or other indicators of significant cognitive impairment or psychiatric disturbance that, in the PI's judgment, precludes participation; and currently receiving cognitive-behavioral therapy.

  * Participants will be invited to complete assessments of salivary cortisol and/or EEG as part of Phase 4, Part 3 study activities. Those who decline completion of these assessments will still be eligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rare and Breast cancer survivors will be recruited to the study. There are no physical recruitment sites outside of MSKCC. Participants may be patients who were treated at MSKCC or rare or breast cancer survivors who were treated elsewhere and learned about the study through an advertisement. The study summary and research team contact information will be available/advertised in the community through MSKCC Connections, MSKCC Survivorship Program and the American Cancer Society website.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2012-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Develop and refine materials (iThrive and iTrack) | 1 year
  This will involve development of a mobile app-based intervention program (based on our results from Phase 1 and 2 and preliminary work conducted by Beard et al.) that targets fear of cancer recurrence for breast, rare gynecological, rare melanoma and skin, long-term adult pediatric, and other rare cancer survivors.

SECONDARY OUTCOMES:
Determine feasibility, usability, acceptability | 1 year
  We will evaluate three versions of the app-based intervention program (iThrive 8, iThrive 16, and iTrack) in BCS (n=30) and RCS (n=90). This will allow us to assess the feasibility of the research procedures, the appropriateness of the psychological and physiological outcome measures, preliminary estimates of pre- and post-intervention effect sizes and reliable change estimates, and variables associated with any observed outcomes.
Preliminary Efficacy | 1 year
  We will evaluate three versions of the app-based intervention program (iThrive 8, iThrive 16, and iTrack) in BCS (n=30) and RCS (n=90). This will allow us to assess the feasibility of the research procedures, the appropriateness of the psychological and physiological outcome measures, preliminary estimates of pre- and post-intervention effect sizes and reliable change estimates, and variables associated with any observed outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT01517945/ICF_000.pdf